CLINICAL TRIAL: NCT00936715
Title: A Rollover Protocol to Provide Open-Label Emtricitabine/Tenofovir Disoproxil Fumarate Combination Product to Subjects Completing the GS-US-203-0107 Study
Brief Title: Rollover Protocol Continued Access to Emtricitabine/Tenofovir Disoproxil Fumarate for Adults in United States
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-203-0109
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Chronic Hepatitis B
Keywords: prevention of chronic hepatitis B recurrence; post orthotopic liver transplant; prevention of chronic hepatitis B recurrence in patients who have undergone orthotopic liver transplant
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- FTC/TDF (Experimental)
  Interventions: Drug: FTC/TDF

INTERVENTIONS:
Drug: FTC/TDF — 200/300 mg tablet administered orally once daily
  Other Names: Truvada®

SUMMARY:
The objective of this study is to provide open label emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) for an additional 5 years (240 weeks) to adults completing study GS-US-203-0107.

ELIGIBILITY:
Key Inclusion Criteria:

* Complete all end of study visit procedures and pharmacokinetic (PK) substudy (if applicable) for the GS US 203 0107 study.
* A negative pregnancy test is required for female individuals at the end of study visit for GS US 203 0107 (unless surgically sterile or greater than two years post-menopausal).
* All sexually active female individuals who are not post menopausal, or surgically sterile and are of childbearing potential must agree to use a highly effective method of contraception during heterosexual intercourse throughout the study.
* Male individuals who are sexually active are required to use barrier contraception (condom with spermicide) during heterosexual intercourse through to study completion.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (4):
- United States (4):
  - Los Angeles, California
  - San Francisco, California
  - Miami, Florida
  - New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the US. The first participant was screened on 06 Aug 2009. The last study visit occurred on 20 November 2015.
Pre-assignment Details: 51 participants were screened.
Groups:
- FTC/TDF: Emtricitabine/tenofovir disoproxil fumarate (FTC/TDF, Truvada®) (200/300 mg) fixed dose combination (FDC) tablet administered once daily for up to 240 weeks.
Period: Overall Study
Arm/Group | FTC/TDF
Started | 24
Completed | 18
Not Completed | 6
Not completed — Investigators Discretion | 1
Not completed — Protocol Violation | 1
Not completed — Safety or Tolerability Reasons | 4

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: participants who were enrolled into the study and received study drug
Groups:
- FTC/TDF: FTC/TDF (200/300 mg) FDC tablet administered once daily for up to 240 weeks
Arm/Group | FTC/TDF
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (10.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 19
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 12
  Black or American African | 5
  Other | 1
  White | 6
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 3
  Non-Hispanic/Latino | 20
  Not Permitted | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Access to, and Received the Intervention
Description: This endpoint has been included to satisfy the requirements of ClinicalTrials.gov. However, there were no prespecified endpoints in this study.
Time Frame: Up to 240 weeks
Population: Participants who were enrolled into the study and received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | FTC/TDF
Number analyzed (Participants) | 24
Participants | 24

ADVERSE EVENTS:
Time Frame: Up to 240 weeks plus 30 days
Description: Non serious/other adverse events were not collected per study protocol.
Groups:
- FTC/TDF: FTC/TDF (200/300 mg) FDC tablet administered orally once daily for up to 240 weeks
Arm/Group | FTC/TDF
Serious Adverse Events (participants affected / at risk) | 7/24
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FTC/TDF (N=24)
Bile duct obstruction Hepatobiliary disorders (Hepatobiliary disorders) | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bipolar disorder (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Appendicectomy (Surgical and medical procedures) | 1
Lung lobectomy (Surgical and medical procedures) | 1
Blood pressure inadequately controlled (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years